CLINICAL TRIAL: NCT00483574
Title: Safety Study of Menactra® (Meningococcal [Groups A, C, Y and W-135] Polysaccharide Diphtheria Toxoid Conjugate Vaccine) When Administered With Other Pediatric Vaccines to Healthy Toddlers
Brief Title: Study of the Safety of Menactra® Vaccine When Administered With Other Pediatric Vaccines to Healthy Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA48
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Meningococcal Meningitis; Measles; Mumps; Rubella; Varicella
Keywords: Menactra® vaccine; Meningococcal meningitis; Measles; Mumps; Rubella; Varicella virus; Haemophilus influenzae type b; Pneumococcal conjugate vaccine
MeSH Terms: conditions — Meningitis, Meningococcal; Measles; Mumps; Rubella; Chickenpox; Haemophilus Infections | interventions — Meningococcal Vaccines; measles, mumps, rubella, varicella vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Menactra® and Routine Pediatric Vaccines (Experimental): Participants received Menactra® alone at age 9 months and Menactra® concomitantly with routine pediatric vaccines (measles-mumps-rubella-varicella [MMRV: ProQuad], pneumococcal conjugate [PCV], and hepatitis A [HepA]) at age 12 months.
  Interventions: Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate; Biological: Measles-mumps-rubella-varicella vaccine; Biological: Routine paediatric vaccine - Pneumococcal conjugate (PCV); Biological: Routine paediatric vaccine - Hepatitis A
- Group 2: Routine Pediatric Vaccines (Other): Participants received routine pediatric vaccines (measles-mumps-rubella-varicella [MMRV: ProQuad], pneumococcal conjugate[PCV], and hepatitis A [HepA]) at age 12 months.
  Interventions: Biological: Measles-mumps-rubella-varicella vaccine; Biological: Routine paediatric vaccine - Pneumococcal conjugate (PCV); Biological: Routine paediatric vaccine - Hepatitis A

INTERVENTIONS:
Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, IM at age 9 and 12 months
  Other Names: Menactra®
  Arms: Group 1: Menactra® and Routine Pediatric Vaccines
Biological: Measles-mumps-rubella-varicella vaccine — 0.5 mL, intramuscular at 12 months of age
  Other Names: MMRV: ProQuad
Biological: Routine paediatric vaccine - Pneumococcal conjugate (PCV) — 0.5 mL, Intramuscular at age 12 months
  Other Names: Pneumococcal conjugate (PCV),
Biological: Routine paediatric vaccine - Hepatitis A — 0.5 mL, Intramuscular at age 12 months
  Other Names: Hepatitis A

SUMMARY:
This clinical trial will evaluate the safety of two injections of Menactra® Vaccine in subjects at 9 months and at 12 months of age when the second dose is given concomitantly with other pediatric vaccines routinely administered in the US.

Safety Objective:

To describe the safety profile of two doses of Menactra® Vaccine.

ELIGIBILITY:
Inclusion Criteria :

* Healthy, as determined by medical history and physical examination
* Aged 9 months (249 to 305 days) or 12 months (365 to 400 days) at the time of enrollment
* The parent or legal guardian has signed and dated the Independent Ethics Committee (IEC)-/Institutional Review Board (IRB)-approved informed consent form.

Exclusion Criteria :

* Serious acute or chronic disease (e.g., cardiac, renal, metabolic, rheumatologic, psychiatric, hematologic, autoimmune disorders, diabetes, atopic conditions, congenital defects, convulsions, encephalopathy, blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic system, acute untreated tuberculosis) that could interfere with trial conduct or completion.
* Known or suspected impairment of immunologic function.
* Acute medical illness within the last 72 hours or a temperature ≥ 100.4ºF (≥ 38.0ºC) at the time of enrollment.
* History of documented invasive meningococcal disease or previous meningococcal vaccination.
* Has received the fourth dose of Prevnar, or the first dose of measles-mumps-rubella (MMR), varicella, or hepatitis A (HepA) vaccine.
* Known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C seropositivity as reported by the parent or legal guardian.
* Received either immune globulin or other blood products within the last 3 months.
* Suspected or known hypersensitivity to any of the vaccine components.
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular (IM) vaccination.
* Parent or legal guardian unable or unwilling to comply with the study procedures.
* Participation in another interventional clinical trial in the 30 days preceding enrollment, or participation in another clinical trial involving the investigation of a drug, vaccine, medical procedure, or medical device during the subject's trial period.
* Diagnosed with any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* Received any vaccine in the 30-day period prior to receipt of the study vaccine(s), or scheduled to receive any vaccination other than influenza vaccination and hyposensitization therapy in the 30-day period after receipt of the study vaccine(s).
* Personal or family history of Guillain-Barré Syndrome (GBS).
* History of seizures, including febrile seizures, or any other neurologic disorder.
* Known hypersensitivity to dry natural rubber latex.

For the subjects scheduled to provide blood samples:

- Anticipated to receive oral or injected antibiotic therapy within the 72 hours prior to either of the study blood draws. Topical antibiotics and antibiotic drops are not included in this exclusion criterion.

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1378 (Actual)
Dates: Start 2007-05; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (72):
- United States (71):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Pinson, Alabama
  - Tuscaloosa, Alabama
  - Chandler, Arizona
  - Bentonville, Arkansas
  - Conway, Arkansas
  - Hardy, Arkansas
  - Jonesboro, Arkansas
  - Downy, California
  - Fountain Valley, California
  - Huntington Beach, California
  - Huntington Park, California
  - La Jolla, California
  - LaCosta, California
  - Pico Rivera, California
  - Centennial, Colorado
  - Longmont, Colorado
  - Thornton, Colorado
  - Lake Mary, Florida
  - Tampa, Florida
  - Stone Mountain, Georgia
  - Boise, Idaho
  - Evansville, Indiana
  - Arkansas City, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Fall River, Massachusetts
  - Clifton, New Jersey
  - Endwell, New York
  - Liverpool, New York
  - Utica, New York
  - Garner, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Minot, North Dakota
  - Cincinnati, Ohio
  - Fairfield, Ohio
  - Huber Heights, Ohio
  - Kettering, Ohio
  - Mason, Ohio
  - Poland, Ohio
  - Youngstown, Ohio
  - Meadowbrook, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Barrington, Rhode Island
  - Providence, Rhode Island
  - Warwick, Rhode Island
  - Barnwell, South Carolina
  - Mt. Pleasant, South Carolina
  - Watertown, South Dakota
  - Bristol, Tennessee
  - Jackson, Tennessee
  - Tullahoma, Tennessee
  - Amarillo, Texas
  - Carrollton, Texas
  - Fort Worth, Texas
  - Grapevine, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - West Valley City, Utah
  - Newport News, Virginia
  - Norfolk, Virginia
  - Vienna, Virginia
  - Bellingham, Washington
- Santiago, Chile

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 30 May 2007 to 28 March 2008 at 82 US clinical centers.
Pre-assignment Details: A total of 1378 participants met inclusion and exclusion criteria, of which 1374 were vaccinated and included in this analysis.
Groups:
- Group 1: Menactra and Routine Pediatric Vaccines: Participants received Menactra alone at age 9 months and Menactra concomitantly with routine pediatric vaccines Measles, mumps and rubella (MMR: M-M-R®II) and varicella (V: Varivax), (0.5 mL Subcutaneous, respectively); pneumococcal conjugate (PCV), and hepatitis A (HepA) at age 12 months. (0.5 mL, intramuscular, respectively)
- Group 2: Routine Pediatric Vaccines: Participants received routine pediatric vaccines, Measles, mumps and rubella (MMR: M-M-R®II) and varicella (V: Varivax), (0.5 mL Subcutaneous, respectively); pneumococcal conjugate (PCV), and hepatitis A (HepA) at age 12 months. (0.5 mL, intramuscular, respectively)
Period: Overall Study
Arm/Group | Group 1: Menactra and Routine Pediatric Vaccines | Group 2: Routine Pediatric Vaccines
Started | 1053 | 321
Completed | 951 | 308
Not Completed | 102 | 13
Not completed — Adverse Event | 6 | 0
Not completed — Protocol Violation | 28 | 9
Not completed — Lost to Follow-up | 16 | 4
Not completed — Withdrawal by Subject | 52 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Menactra and Routine Pediatric Vaccines | Group 2: Routine Pediatric Vaccines | Total
Number analyzed (Participants) | 1053 | 321 | 1374
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1053 | 321 | 1374
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 282.8 (10.79) | 374.6 (8.93) | 304.3 (40.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 511 | 158 | 669
  Male | 542 | 163 | 705
Region of Enrollment [Number; unit: participants]
  United States | 1053 | 321 | 1374

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Solicited Injection Site Reaction or Systemic Reaction Following Vaccination.
Description: Solicited injection site reactions: tenderness, Erythema (Redness), and Swelling.
  Solicited systemic reactions: Fever (Temperature), Vomiting, Crying Abnormal, Drowsiness, Appetite Lost, and Irritability
Time Frame: Day 0 to 7 Post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population. Data on 23 participants in Group 1 that received MMR+V vaccines instead of a MMRV single vaccine in addition to the PCV and HepA vaccines were analyzed separately.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Menactra and Routine Pediatric Vaccines | Group 2: Routine Pediatric Vaccines
Number analyzed (Participants) | 1030 | 321
Percentage of participants
  Any Injection Site Reaction at 9 Months - Menactra | 52 | NA — Participants did not receive Menactra vaccine
  Any Tenderness at 9 Months - Menactra | 37 | NA — Participants did not receive Menactra vaccine
  Grade 3 Tenderness (Cries when limb is moved) | 1 | NA — Participants did not receive Menactra vaccine
  Any Erythema at 9 Months - Menactra | 30 | NA — Participants did not receive Menactra vaccine
  Grade 3 Erythema (≥ 2.0 in [≥ 5.0 cm]) | 0 | NA — Participants did not receive Menactra vaccine
  Any Swelling at 9 Months - Menactra | 17 | NA — Participants did not receive Menactra vaccine
  Grade 3 Swelling (≥ 2.0 in [≥ 5.0 cm]) | 0 | NA — Participants did not receive Menactra vaccine
  Any Injection Site Reaction at 12 Months -Menactra | 58 | NA — Participants did not receive Menactra vaccine
  Any Tenderness at 12 Months - Menactra | 49 | NA — Participants did not receive Menactra vaccine
  Grade 3 Tenderness (Cries when limb is moved) | 1 | NA — Participants did not receive Menactra vaccine
  Any Erythema at 12 Months - Menactra | 30 | NA — Participants did not receive Menactra vaccine
  Grade 3 Erythema (≥ 2.0 in [≥ 5.0 cm]) | 0 | NA — Participants did not receive Menactra vaccine
  Any Swelling at 12 Months - Menactra | 16 | NA — Participants did not receive Menactra vaccine
  Grade 3 Swelling (≥ 2.0 in [≥ 5.0 cm]) | 0 | NA — Participants did not receive Menactra vaccine
  Any Injection Site Reaction at 12 Months, MMRV | 44 | 59
  Any Tenderness at 12 Months - MMRV | 39 | 43
  Grade 3 Tenderness (Cries when limb is moved) | 1 | 0
  Any Erythema at 12 Months - MMRV | 23 | 33
  Grade 3 Erythema (≥ 2.0 in [≥ 5.0 cm]) | 0 | 0
  Any Swelling at 12 Months - MMRV | 12 | 14
  Grade 3 Swelling (≥ 2.0 in [≥ 5.0 cm]) | 0 | 0
  Any Injection Site Reaction at 12 Months, PCV | 53 | 56
  Any Tenderness at 12 Months - PCV | 46 | 46
  Grade 3 Tenderness (Cries when limb is moved) | 2 | 0
  Any Erythema at 12 Months - PCV | 29 | 33
  Grade 3 Erythema (≥ 2.0 in [≥ 5.0 cm]) | 0 | 1
  Any Swelling at 12 Months - PCV | 20 | 17
  Grade 3 Swelling (≥ 2.0 in [≥ 5.0 cm]) | 0 | 1
  Any Injection Site Reaction at 12 Months, HepA | 50 | 52
  Any Tenderness at 12 Months - HepA | 43 | 41
  Grade 3 Tenderness (Cries when limb is moved) | 1 | 0
  Any Erythema at 12 Months - HepA | 25 | 27
  Grade 3 Erythema (≥ 2.0 in [≥ 5.0 cm]) | 0 | 0
  Any Swelling at 12 Months - HepA | 16 | 14
  Grade 3 Swelling (≥ 2.0 in [≥ 5.0 cm]) | 0 | 0
  Any Systemic Reaction at 9 Months | 69 | 0
  Any Fever, (rectal or oral temperature route) | 12 | 0
  Grade 3 Fever (>103.1 ºF [>39.5 ºC]), Any Route | 1 | 0
  Any Vomiting at 9 Months | 14 | 0
  Grade 3 Vomiting (≥ 6 episodes per 24 hours) | 0 | 0
  Any Crying Abnormal at 9 Months | 33 | 0
  Grade 3 Crying Abnormal (> 3 hours) | 2 | 0
  Any Drowsiness at 9 Months | 30 | 0
  Grade 3 Drowsiness (Sleeps most of time) | 1 | 0
  Any Appetite Lost at 9 Months | 30 | 0
  Grade 3 Appetite Lost (Refuses ≥ 3 feeds/meals) | 1 | 0
  Any Irritability at 9 Months | 57 | 0
  Grade 3 Irritability (Inconsolable) | 3 | 0
  Any Solicited Systemic Reaction at 12 Months | 73 | 75
  Any Fever, (rectal or oral temperature route) | 25 | 22
  Grade 3 Fever (>103.1 ºF [>39.5 ºC]), Any Route | 2 | 3
  Any Vomiting at 12 Months | 11 | 10
  Grade 3 Vomiting (≥ 6 episodes per 24 hours) | 0 | 0
  Any Crying Abnormal at 12 Months | 40 | 39
  Grade 3 Crying Abnormal (> 3 hours) | 2 | 1
  Any Drowsiness at 12 Months | 40 | 39
  Grade 3 Drowsiness (Sleeps most of time) | 1 | 1
  Any Appetite Lost at 12 Months | 36 | 32
  Grade 3 Appetite Lost (Refuses ≥ 3 feeds/meals) | 3 | 1
  Any Irritability at 12 Months | 62 | 65
  Grade 3 Irritability (Inconsolable) | 4 | 4

2. Other Pre Specified Outcome: Safety Overview After Any Vaccination in Participants Who Received MMR+V
Time Frame: Day 0 to 7 Post-vaccination
Population: Summary of the safety analysis of the 23 participants in Group 1 that received MMR+V vaccines instead of a MMRV single vaccine in addition to the PCV and HepA vaccines.
Measure: Number; unit: Percentage of participants
Groups:
- Group 1: Menactra and Routine Pediatric Vaccines: Participants received Menactra alone at age 9 months and Menactra concomitantly with routine pediatric vaccines (measles-mumps-rubella-varicella [MMR+V: ProQuad], pneumococcal conjugate [PCV], and hepatitis A [HepA]) at age 12 months. (0.5 mL, intramuscular, respectively)
Arm/Group | Group 1: Menactra and Routine Pediatric Vaccines | Group 2: Routine Pediatric Vaccines
Number analyzed (Participants) | 23 | 0
Percentage of participants
  Injection Site Reaction at 9-Month, Menactra | 44 |
  Injection Site Reaction at 12-Month, Menactra | 57 |
  Injection Site Reaction at 12-Month, MMR | 52 |
  Injection Site Reaction at 12-Month, Varivax | 41 |
  Injection Site Reaction at 12-Month, PCV | 68 |
  Injection Site Reaction at 12-Month, HepA | 65 |
  Any Solicited Systemic Reaction at 9-Month vac | 52 |
  Any Solicited Systemic Reaction at 12-Month vac | 70 |
  Unsolicited Adverse Event at 9-Month | 52 |
  Unsolicited Adverse Event at 12-Month | 36 |
  Serious Adverse Events | 0 |

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for up to 6 months after the last vaccination.
Arm/Group | Group 1: Menactra and Routine Pediatric Vaccines | Group 2: Routine Pediatric Vaccines
Serious Adverse Events (participants affected / at risk) | 42/1053 | 5/321
Other Adverse Events (participants affected / at risk) | 530/1053 | 95/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Menactra and Routine Pediatric Vaccines (N=1053) | Group 2: Routine Pediatric Vaccines (N=321)
Inborn error of metabolism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 5 (6) | 0 (0)
Campylobacter intestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Croup Infections (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Febrile convulsion (Nervous system disorders) | 7 (8) | 0 (0)
Breath holding (Psychiatric disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Bronchial hyperactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Menactra and Routine Pediatric Vaccines (N=1053) | Group 2: Routine Pediatric Vaccines (N=321)
Diarrhoea (Gastrointestinal disorders) | 109 (126) | 18 (20)
Injection site bruising (General disorders) | 85 (102) | 18 (20)
Pyrexia (General disorders) | 65 (76) | 17 (18)
Otitis media (Infections and infestations) | 183 (210) | 26 (27)
Upper respiratory tract infection (Infections and infestations) | 150 (165) | 16 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 133 (146) | 13 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 82 (90) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 53 (55) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.